CLINICAL TRIAL: NCT05770622
Title: The VANcomycin Cohort Study - Assessing Precise Dosing and Prompt Drug Monitoring to Improve Attainment of Target Concentrations (Part 2)
Brief Title: Improving Therapeutic Drug Monitoring and Dosing for Vancomycin in Young Infants With Infections (VANCAPP) (Part 2)
Acronym: VANCAPP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Royal Children's Hospital (Other); Royal Hospital For Women (Other); Sydney Children's Hospitals Network (Other); Monash Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HREC2019.059 (part 2)
Record Dates: First submitted 2023-03-05; First posted 2023-03-15 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-06

CONDITIONS: Sepsis; Infections; Bacteremia
MeSH Terms: conditions — Sepsis; Infections; Bacteremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vancomycin first-dose trough dose adjustment calculation (Experimental): Participants will have individualised model-based intermittent vancomycin dosing using the Vanc App dosing calculator (as used in VANC APP Part 1, see clinicaltrials.gov ID: NCT04044703). A first-dose trough concentration will be measured for each participant and the clinician will then enter that concentration into the web application ('First-dose trough dose adjustment calculator'). A dose adjustment will be generated by the calculator if the predicted steady-state level is outside of target range. If the predicted steady-state level is within target range (10-20mg/L) the calculator will recommend continuing with the same dose. The vancomycin concentration is then measured at steady state to determine if the target concentration has been achieved.
  Interventions: Other: First-dose trough dose adjustment calculator - using early TDM (first-dose trough) to determine an early dose adjustment if the predicted steady-state trough is outside of target range (10-20mg/L)

INTERVENTIONS:
Other: First-dose trough dose adjustment calculator - using early TDM (first-dose trough) to determine an early dose adjustment if the predicted steady-state trough is outside of target range (10-20mg/L) — CALCULATOR: A 'First-dose trough dose adjustment calculator' was developed based on a population pharmacokinetic model. A participant's post-menstrual age, weight, creatinine, target trough concentration, dose, dosing interval and first-dose trough concentration (taken immediately before the second dose is due) are entered into the calculator. The calculator determines if a dose adjustment is required (based on whether the predicted steady-state trough concentration is <10mg/L or >20mg/L) and, if required, recommends a new adjusted dose.

SUMMARY:
A challenge to intermittent vancomycin dosing in young infants is the avoidable delay caused by the need to wait until steady state (i.e. when the drug concentrations are in equilibrium) to measure a vancomycin concentration, as this generally occurs 24 to 48 hours after starting treatment. If the target concentration is not achieved, the dose needs to be adjusted, resulting in further delays in an infant achieving the concentration required to treat their infection. The purpose of this study is to assess the use of early therapeutic drug monitoring (first-dose trough) and, if needed, early dose adjustment, in achieving target vancomycin concentrations at steady state. A dose adjustment calculator (available through a web application) will be used to determine the need for dose adjustment (based on predicted steady state concentration) and recommend an adjusted dose if required.

DETAILED DESCRIPTION:
Therapeutic drug monitoring (TDM) for vancomycin is done once the drug is in steady state. In young infants, this occurs at 24-48hours after commencing vancomycin. If the concentration at steady state is not in therapeutic range (10-20 mg/L), the dose is adjusted and the concentration measured again 24 hour later. Using empiric vancomycin dosing regimens, fewer than 50% of infants achieve the target concentration at their first steady state level. Therefore once the dose is adjusted and concentration repeated, there is a delay of at least 48 hours before adequate antibiotic concentrations are achieved in the blood - delaying optimal treatment of life-threatening infections. This study aims to use early TDM and dose adjustment to improve the proportion of infants achieving target concentrations at their first steady-state level.

Using a published population pharmacokinetic model, we identified a linear relationship between the first-dose trough and steady-state trough (R2 = 0.51) as well as the first-dose trough and AUC24 at 48 hours (R2= 0.70). This suggests that TDM could be performed after the first dose and that this early trough level could be used to predict the steady state level, enabling earlier dose adjustment and thereby shortening the time to effective therapy. This model has therefore been used to develop an online 'First-dose trough dose adjustment calculator'.

In the VANC APP (Part 2)* study, participants will have individualised model-based intermittent vancomycin dosing using the Vanc App dosing calculator (as used in VANC APP Part 1, see clinicaltrials.gov ID: NCT04044703). A first-dose trough concentration will be measured for each participant and the clinician will then enter that concentration into the web application ('First-dose trough dose adjustment calculator'). A dose adjustment will be generated by the calculator if the predicted steady-state level is outside of target range. The vancomycin concentration is then measured at steady state to determine if the target concentration has been achieved.

*Note: This study is 'part 2' of the VANC APP study protocol as approved under HREC reference number HREC/51942/RCHM-2019. Part 1 was registered separately on clinicaltrials.gov (clinicaltrials.gov ID: NCT04044703). Part 1 has been completed and assessed the use of model-based individualised intermittent vancomycin dosing using the Vanc App dosing calculator in 40 young infants aged 0 to 90 days. The vancomycin concentration was measured at steady state (24-48 hours) to determine the proportion of infants achieving target concentrations. Part 1 and part 2 are two separate studies and the results of each part will not be directly compared to one another.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 0 - 90 days old
* Suspected infection requiring treatment with vancomycin for 48 hours or more (as determined by the clinical team)

Exclusion Criteria:

* Infants with a corrected gestational age of less than 25 weeks
* Infants weighing less than 500g.
* Known allergy to any glycopeptide antibiotic
* Vancomycin administered within the previous 72 hours
* Infants receiving any form of extracorporeal life support
* Renal impairment

Ages: 0 Days to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Target concentration at first steady-state concentration | From first vancomycin dose (immediately after consent) to steady state level taken at 24-48 hours post-first-dose
  The proportion of young infants achieving target trough serum vancomycin concentrations (10 to 20 mg/L) at first steady-state level when model-based dosing is used followed by early therapeutic drug monitoring (and dose adjustment) after the first dose

SECONDARY OUTCOMES:
Sub- and supratherapeutic concentrations at first steady-state concentration | From first vancomycin dose (immediately after consent) to steady state level taken at 24-48 hours post-first-dose
  The proportion of young infants with supra- (defined as >20mg/L) or sub- (defined as <10mg/L) therapeutic vancomycin concentrations at the first steady state level when model-based dosing is used followed by early therapeutic drug monitoring (and dose adjustment) after the first dose
Drug-related adverse effects | From first vancomycin dose (immediately after consent) to completion of vancomycin therapy (as determined by clinical team, an average of 5 days)
  The frequency of drug-related adverse effects (infusion-related and nephrotoxicity).

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Wilkins, MBBS, Principal Investigator — Royal Children's Hospital Melbourne, Murdoch Children's Research Institute
Locations (4):
- Australia (4):
  - Royal Children's Hospital Melbourne, Melbourne, Victoria
  - Monash Newborn, Melbourne
  - Royal Hospital for Women, Sydney
  - The Children's Hospital at Westmead, Sydney

IPD SHARING:
Plan to Share IPD: No